CLINICAL TRIAL: NCT05043051
Title: Autoimmune Basis for Postural Tachycardia Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 13705; 2R01HL128393-04 (NIH)
Record Dates: First submitted 2021-08-27; First posted 2021-09-13 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Postural Tachycardia Syndrome
Keywords: POTS; Vagal Stimulation; Autoantibody
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Vagus Nerve Stimulation; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vagal stimulation (Active Comparator): Vagal stimulation will be given at 20 Hz for 1 hour daily with the bipolar electrode attached to the tragus for 2 months.
  Interventions: Device: Vagal stimulation
- Sham stimulation (Sham Comparator): Sham stimulation will be given at 20 Hz for 1 hour daily with the bipolar electrode attached to the earlobe for 2 months.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Vagal stimulation — Vagal stimulation
  Other Names: Transcutaneous electrical nerve stimulation
  Arms: Vagal stimulation
Device: Sham stimulation — Sham vagal stimulation
  Other Names: Transcutaneous electrical nerve stimulation
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is to test the hypothesis that an antibody-mediated autoimmune reaction will cause symptoms of autonomic dysfunction in some patients with postural tachycardia syndrome (POTS). The investigators further hypothesize that electrical stimulation of the vagus nerve will improve POTS symptoms, autoimmunity and inflammation.

DETAILED DESCRIPTION:
The present study is designed to test the hypothesis that muscarinic autoantibody-mediated parasympathetic dysfunction contributes to the pathogenesis of POTS, and that parasympathetic (vagal) stimulation improves POTS symptoms, autoimmunity and inflammation.

Define and determine the prevalence, burden, and clinical significance of muscarinic autoantibodies in a well-phenotyped cohort of POTS patients with and without gastroparesis and a matched cohort of healthy control subjects.

Evaluate the impact of vagal stimulation on antibody suppression, inflammatory inhibition, and symptom improvement in POTS patients. Non-invasive transcutaneous stimulation of the auricular branch of the vagus nerve (tragus stimulation) will be used to increase parasympathetic activity.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old, female or male
* Either healthy control or individual with postural tachycardia syndrome (POTS) defined as heart rate increase >30 bpm from supine within 10 min of standing, in the absence of orthostatic hypotension (>20/10 mmHg fall in blood pressure), with chronic symptoms (>6 months), and in the absence of other acute cause of orthostatic tachycardia
* Able and willing to provide informed consent
* Understand and be able to comply with the study procedures and restrictions

Exclusion Criteria:

* Hypertension (>150 mmHg systolic and >100 mmHg diastolic) based on history or findings at screening
* Orthostatic hypotension (consistent drop in blood pressure >20/10 mmHg with 10 min of standing)
* Cardiovascular disease, such as myocardial infarction within 6 months
* History or presence of significant immunological or hematological disorders
* History of vagotomy
* Currently pregnant women or women planning on becoming pregnant ≤ 3 months
* Inability to comply with the protocol
* Patients with active implants (such as a cardiac pacemaker, or a cochlear implant)

Healthy control subjects will be healthy, non-smoking and on no chronic medications at the time of the study. Healthy control subjects will be group-matched to the POTS patients for age and gender.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 5 minute
  Average of heart rate variability during the posture test

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Stavrakis, MD, Study Director — University of Oklahoma
Locations (1):
- Oklahoma Clinical and Translational Science Institute, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stavrakis S, Chakraborty P, Farhat K, Whyte S, Morris L, Abideen Asad ZU, Karfonta B, Anjum J, Matlock HG, Cai X, Yu X. Noninvasive Vagus Nerve Stimulation in Postural Tachycardia Syndrome: A Randomized Clinical Trial. JACC Clin Electrophysiol. 2024 Feb;10(2):346-355. doi: 10.1016/j.jacep.2023.10.015. Epub 2023 Nov 22. PMID 37999672